CLINICAL TRIAL: NCT05308849
Title: Peritoneal Diffusion and Efficacy of Antibiotic Therapy in Pediatric Peritonitis
Acronym: DIFFUPERPED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: PAPE Elise (Unknown)
Responsible Party: Principal Investigator, Nicolas BERTE, Principal Investigator, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021-A00378-33
Record Dates: First submitted 2022-01-20; First posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Peritonitis; Appendicitis; Children, Only; Antibiotic Toxicity
Keywords: Children Peritonitis; Antibiotic diffusion; Pharmacocinetic study
MeSH Terms: conditions — Peritonitis; Appendicitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pediatric Peritonitis (Other): Patient (from 3 to 17 years-old) treated for appendicular peritonitis. It includes surgical treatment (appendicectomy, peritoneal toilet) and antibiotherapy according to French recommendation.
  Interventions: Other: Dosage of serum and peritoneal of the betalactam used for antibiotic treatment

INTERVENTIONS:
Other: Dosage of serum and peritoneal of the betalactam used for antibiotic treatment — All patients will have antibiotherapy according to French recommendation.
  Antibiotics recommended are:
  cefotaxime 200mg/kg/d / OR amoxicillin/clavulanic acid 25 mg/kg x 3 /d OR piperacilline/tazobactam 100 mg/kg/d
  Blood samples will be collected before surgery and after surgery (for all patients).
  Peritoneal sample will be collected during surgery (for all patients). Additionnal optionnal blood sample could be collected on Day 5 after surgery. Additionnal optionnal peritoneal samples could be collected on Day 2 and Day 5.
  Dosage of serum and peritoneal of the used betalactam will be performed by High Performance Liquid Chromatography Method

SUMMARY:
This is a pilote monocentric prospective study about pediatric peritonitis and antibiotics pharmacokinetic and pharmacodynamic. The investigators will include 41 patients between 3 and 17 years-old during 2 years in the University Hospital of Nancy.

The aim of this study is to determine if the beta-lactam dosages in children recommended by the guidelines for management of intra-abdominal infections permitted the achievement of adequatly serum and peritoneal concentrations in the medical and surgical management of peritonitis.

The investigators will collected serum and peritoneal fluid samples at 3 different times: peritoneal incision, end of surgery, 2 days and 5 days after surgery in order to compare the concentrations and the minimal inhibitor concentration of bacteria.

The hypothesis is that of a serum and peritoneal antibiotic under dosage.

DETAILED DESCRIPTION:
Pediatric population with localized or generalized appendicular peritonitis with surgical management at the Nancy University Hospital.

Patients are usually taken in emergency at the Pediatric Emergency Department (Children's Hospital, CHRU Nancy). The diagnosis of peritonitis is then made or confirmed by clinical examination and paraclinical tests (biology and imaging).

Written informed consent is obtained from one of the parental authority holders, allowing inclusion in the study. An information document adapted to the child's understanding will also be sent to him/her. The child's non-opposition will be sought if he/she is old enough to understand. The information will be given jointly to the child and to the legal guardians present at the patient's bed at the time of diagnosis of peritonitis. The reflection period will correspond to the interval between this information and the management in the operating room. This may vary depending on the occupation of the operating room.

The diagnosis of appendicular peritonitis is made by the surgeon (routine care). The child is included.

Antibiotic therapy is started IV according to the protocol in force at the CHRU (routine care):

- Cefotaxime (200 mg/kg/d, 4 IV administrations) + Metronidazole (20-30 mg/kg/d, 3 IV administrations)+/-Gentamicin (3-8 mg/kg/d IV)

Specific biological samples and collections are taken for the research:

* A blood sample (1mL) (S0) after injection of the antibiotic and before appendicular section, non-invasive because performed on peripheral venous route.
* A blood sample (1mL) (S1) at the end of the operation, either when the peripheral venous route is placed if possible (non-invasive), otherwise at the periphery (invasive).
* If a drainage of the peritoneal cavity is in place, a non-invasive collection of peritoneal fluid (5 mL) on the drain will be performed (P1) at D2.
* If generalized peritonitis, an additional blood collection (1mL) at D5 (S2) during the biological check-up (routine care). If an abdominal drainage is still in place, a non-invasive collection of peritoneal fluid (5mL) on drain will be performed (P2). At D5, the patients are under appropriate antibiotic therapy.

Specifically for research, betalactam assays are performed on S0, S1, S2, P0, P1 and P2 once all samples have been sent to Pharmacology.

Bacteriological analyses are performed on P0 (routine care), P1 and P2 in real time.

The following specific data will be collected: time of first antibiotic administration, time of sampling (S0, S1 and P0), time of surgery start. Data concerning antibiotic therapy (dosage, frequency of administration) will be collected during the entire hospitalization period as well as the time of the other samples if applicable (S2, P1 and P2).

Clinical and biological data are collected, including the visit at 4-6 weeks after discharge. (In routine care, a visit at 1 month post-op is performed). The investigator looks for AEs or SAEs. At the end of this post-operative visit, the patient is discharged from the study.

The volume of blood collected in the framework of the research is estimated at 3mL, i.e. less than 2.5% of the total blood volume over the inclusion period. The maximum total volume collected is 24 mL (6 mL for research, 18 mL for care, i.e. 3 samples of CBC, blood ionogram and CRP).

Blood and peritoneal samples :

The 3 blood samples as well as the 2 (possibly 3) peritoneal samples will be taken by a nurse and will be placed in a specific bag. Each sampling time will be clearly identified on the sample and a traceability form will be completed and sent to the Pharmacology and Toxicology laboratory.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of intra-abdominal infection : localized or generalized peritonitis secondary to appendix

Exclusion Criteria:

* betalactams allergy
* peritonitis with other etiology than appendix
* antibiotic treatment longer than 24h

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Estimated)
Dates: Start 2022-03-31 (Estimated); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
antibiotic concentration | Peritoneal incision, end of surgery, Day+5 after surgery if systemic peritonitis,
  Serum betalactams concentrations at different times
antibiotic concentration | During surgery, Day+2 after surgery if drain peritonal, Day+5 after surgery if systemic peritonitis,
  Peritonal betalactams concentrations at different times

SECONDARY OUTCOMES:
Determine elimination rate constant Kel | Statistical analysis after 2 years of inclusion
  It is the first order rate constant describing drug elimination from the body.
Determine estimated initial concentrationf C0 | Statistical analysis after 2 years of inclusion
  Initial concentration of antibiotic in the body
Determine Area Under the Curve AUC. | Statistical analysis after 2 years of inclusion
  It is the definite integral of a curve that describes the variation of a drug concentration in blood plasma as a function of time.
Determine Half-life | Statistical analysis after 2 years of inclusion
  It is a pharmacokinetic parameter that is defined as the time it takes for the concentration of the drug in the plasma or the total amount in the body to be reduced by 50%.
Determine distribution volume | Statistical analysis after 2 years of inclusion
  It is a pharmacokinetic parameter representing an individual drug's propensity to either remain in the plasma or redistribute to other tissue compartments.
Determine Clearance or betalactams in children | Statistical analysis after 2 years of inclusion
  It is a pharmacokinetic measurement of the volume of plasma from which a substance is completely removed per unit time.
Evaluate the relationship between serum and peritoneal concentrations of beta-lactam | Statistical analysis after 2 years of inclusion
  Determination of the antibiotic diffusion coefficient through the peritoneal membrane : difference between serum concentration and peritoneal concentration of betalactam
Proportion of different bacteria | Statistical analysis after 2 years of inclusion
  Describe the local bacterial ecology
Proportion of sensitive and resistant germs to betalactam antibiotics | Statistical analysis after 2 years of inclusion
  Describe the local bacterial ecology
Description of minimal inhibition concentration for bacterias | Statistical analysis after 2 years of inclusion
  Describe the local bacterial ecology
Factors associated with an antibiotic under-dosage | Statistical analysis after 2 years of inclusion
  Factors statistically associated with antibiotic under dosage defined by serum and peritonal concentrations < 4*MIC using multivariate analysis.
Factors associated with an antibiotic overdose | Statistical analysis after 2 years of inclusion
  Factors statistically associated with antibiotic overdose defined by serum and peritonal concentrations >10*MIC using multivariate analysis.
Evaluation of duration of hospitalization | Statistical analysis after 2 years of inclusion
  Describe the clinical efficacy of antibiotic protocol
Mean delay for apyrexia | Statistical analysis after 2 years of inclusion
  Describe the clinical efficacy of antibiotic protocol
Clinical complications | Statistical analysis after 2 years of inclusion
  Describe the clinical efficacy of antibiotic protocol